CLINICAL TRIAL: NCT05476653
Title: A Prospective Monocentric Study to Assess the Concordance of Lung MRI Compared to Chest CT Scan to Assess the Extent and Severity of Bronchial and Parenchymal Pulmonary Lesions in Adult Patients With Primary Immune Deficiency (PID): IRM vs SCANNER
Brief Title: A Prospective Monocentric Study to Assess the Concordance of Lung MRI Compared to Chest CT Scan to Assess the Extent and Severity of Bronchial and Parenchymal Pulmonary Lesions in Adult Patients With Primary Immune Deficiency (PID) .
Acronym: IRMvsSCANNER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Collaborators: Siemens Healthcare QT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021_0015
Record Dates: First submitted 2022-01-31; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Primary Immune Deficiency
Keywords: Primary Immune Deficiency; MRI; Chest CT Scan
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI exam (Experimental): Patients will be asked to perform a pulmonary MRI in addition to the usual chest CT can.
  The chest CT scan will be performed according to the usual protocol of standard practices. No difference is expected for this research protocol.
  Interventions: Other: MRI procedure

INTERVENTIONS:
Other: MRI procedure — Pulmonary MRI based on a 1.5 T machine (Siemens VIDA) or a 3T machine (Siemens SOLA) without the use of contrast product according to a protocol based on a 3D-UTE sequence acquired in free breathing but with a respiratory synchronization system in association with weightings in T1 and T2.

SUMMARY:
Currently, there is no official recommendations for the respiratory surveillance of patients with PID.However, it is recommended to perform a chest CT scan each 5 years or before any significant therapeutic change.

The methods of surveillance need to meet two contradictory imperatives:

* monitor frequently enough not to diagnose with delay an aggravation of bronchiectasis or interstitial pneumonitis, an infectious complication by a slowly growing pathogen such as a non-tuberculous mycobacterium, or lymphoid proliferation.
* do not expose these often young patients to significant irradiation by a considerable number of scans during their life. In addition, some patients with PID have increased radiosensitivity without a safe irradiation threshold having been determined.

To make thoses requirements effective, the solution is to combine radiological monitoring and absence of irradiation. Therefore, it makes sense to study whether chest scans can be replaced by MRI, non-irradiating imaging. But the question that needs to be answered is whether the information provided by the chest MRI is not inferior to that provided by the scanner.

The objective of this study is to assess the ability of MRI performed with ultrashort echo time to analyze the extent and severity of bronchial and pulmonary parenchymal lesions during the follow-up of patients with primary immunodeficiency, comparing them to those of the chest CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Adult patients with PID
* Patients who have performed EFR (Functional Respiratory Tests) within 6 months
* Patients who have signed a consent form
* Patients affiliated with a Health Insurance plan.

Exclusion Criteria:

* Pregnant woman
* Contraindications to MRI:

  * Patients with magnetically activated implanted devices (cardiac pacemakers, insulin pumps, neurostimulators, cochlear implants),
  * Patients with intraocular metal or in the brain (aneurysm clip),
  * Patients with prostheses in the thoracic position and contraindicated for MRI examination
  * Claustrophobic patients.
* To be deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
To assess the bronchial lesions | 6 montths
  Analysis of the presence, the severity (cylindrical, varicose or cystic) and segmental distribution of bronchiectasis, 2. the presence and lobar distribution of hypoperfused pulmonary areas, and 3. the presence and lobar distribution of interstitial abnormality and pulmonary nodular lesions.
  Those three components will be independently identified by lung scanners and MRIs.
To assess the parenchymal lesions | 6 montths
  Analysis of the presence and lobar distribution of hypoperfused pulmonary areas

SECONDARY OUTCOMES:
To assess the MRI results versus the scanner results | 6 months
  To assess the reproducibility of MRI performed using a prototype 3D-UTE SPIRALVIBE sequence and CT scan to detect bronchial and pulmonary parenchymal abnormalities at the segmental, lobar or pulmonary scale, by two independent thoracic radiologists.

CONTACTS AND LOCATIONS:
Overall Officials: 0146252315 Louis-Jean Couderc,MD, Principal Investigator — lj.couderc@hopitalfoch.com
Locations (1):
- Foch hospital, Suresnes, France